CLINICAL TRIAL: NCT01285544
Title: Assessment of the Efficacy and Tolerability of Two Formulations of Atorvastatin In Korean Adult With Hypercholesterolemia : A Multicenter, Prospective, Open-Label, Randomized, Trial
Brief Title: The Efficacy and Tolerability of Two Formulations of Atorvastatin In Korean Adult With Hypercholesterolemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lipinon Study; H-0807-056-251
Record Dates: First submitted 2011-01-09; First posted 2011-01-28 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Dyslipidemia; Cardiovascular Disease; Hypercholesterolemia
Keywords: statins; cholesterol; hypercholesterolemia; atorvastatin; Dyslipidemia in cardiovascular disease (KoLipinon)
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases; Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipinon-test formulation of atrovastain - 20mg (Experimental)
  Interventions: Drug: Atorvastatin (Lipinon)
- Lipitor- branded formuation of atorvastatin-20mg (Active Comparator)
  Interventions: Drug: Atorvastatin (Lipitor)

INTERVENTIONS:
Drug: Atorvastatin (Lipinon) — treatment of dyslipidemia administration : PO, qod
  Arms: Lipinon-test formulation of atrovastain - 20mg
Drug: Atorvastatin (Lipitor) — treatment of dyslipidemia administration : PO, qod
  Arms: Lipitor- branded formuation of atorvastatin-20mg

SUMMARY:
There will be no significant differences in the efficacy and tolerability between the test and reference formulations of atorvastatin 20 mg in these Korean adults with primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* the patients aged 20 to 79 years with primary hypercholesterolemia that was not sufficiently responsive to therapeutic lifestyle changes and had LDL-C level over 100 mg/dL in high risk group.
* Inclusion criteria was in accordance with drug treatment guidelines; coronary artery disease or equivalent group with LDL-C ≥100 mg/dl; patients with two or more risk factors and LDL-C≥130 mg/dl; patients with 0 or 1 risk factor and LDL-C >160 mg/dl after therapeutic lifestyle changes

Exclusion Criteria:

* therapy with any other investigational drug within 30 days of randomization,
* history of hypersensitivity to HMG-CoA reductase inhibitors,
* uncontrolled hypertension,
* poorly controlled diabetes (glycosylated hemoglobin [HbA1c] >9%),
* unstable angina or presented with new-onset myocardial infarction (within 6 months),
* creatinine >2.5 mg/dl,
* alanine aminotransferase (ALT) >2 x upper limit of normal (ULN), aspartate aminotransferase(AST) >2 x ULN, or creatine kinase (CK) >2 x ULN,
* history of malignancy or psychosis;
* chronic liver disease,
* drug or alcohol abuse, pregnancy, breastfeeding, failure to practice adequate contraception, cyclical hormonal contraceptives or intermittent use of hormone replacement therapies.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
the percent change of LDL-C level | After taken medication for 8 weeks

SECONDARY OUTCOMES:
the percent change in total cholesterol, triglyceride, high density lipoprotein cholesterol (HDL-C) level, apolipoprotein B/A1 ratio, LDL/HDL ratio, small dense LDL fraction, high-sensitive C reactive protein (hs-CRP) | After taken medication for 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim SH, Seo MK, Yoon MH, Choi DH, Hong TJ, Kim HS. Assessment of the efficacy and tolerability of 2 formulations of atorvastatin in Korean adults with hypercholesterolemia: a multicenter, prospective, open-label, randomized trial. Clin Ther. 2013 Jan;35(1):77-86. doi: 10.1016/j.clinthera.2012.11.009. Epub 2012 Dec 28. PMID 23274145